CLINICAL TRIAL: NCT03710083
Title: A Pivotal Study to Evaluate Guardian™ Connect CGM System Performance in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP320
Record Dates: First submitted 2018-10-15; First posted 2018-10-17 (Actual); Results first posted 2020-08-21 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Type I Type II
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Study arm (Experimental): Use two Guardian™ Sensor (3)s each connected to a Guardian™ Connect transmitter for approximately 7 days and undergo one Yellow Springs Instrument (YSI™) frequent sample testing (FST) (Day 1, 3-5, or 7).
  Interventions: Device: Guardian™ Sensor (3)

INTERVENTIONS:
Device: Guardian™ Sensor (3) — Use two Guardian™ Sensor (3)s each connected to a Guardian™ Connect transmitter for approximately 7 days.

SUMMARY:
The purpose of this study is to demonstrate the performance and safety of the Guardian™ Sensor (3) over 170 hours (7 days) when inserted in the abdomen used in subjects age 14 - 75 years with the Guardian™ Connect System.

DETAILED DESCRIPTION:
This study is a multi-center, prospective single-arm design without controls. Up to 72 subjects will be enrolled in order to have approximately 60 subjects complete the study. Three investigational centers in China will be used during this study.

During the study, each subject will be randomly assigned to one day of the Yellow Springs Instrument (YSI™*) frequent sample testing (FST) (Day 1, 3-5, or 7).Subjects will wear two Guardian™ Sensor (3)s each connected to a Guardian™ Connect transmitter for approximately 7 days (one which will be paired to the Guardian Connect app and the other will function as a glucose recorder.).

The Guardian Sensor (3)s will be worn in the abdomen area and self-inserted by the subject on same side or opposite sides.

On the evening prior to FST, subjects will be asked to fast for approximately 12 hours and adjust their insulin and medications according to routine care (for example as they would do for fasting lipid panel). Subjects may fast for shorter period of time based on investigator discretion.

The subject should be in fasting status upon arrival hospital to start FST process. The feeding protocol may be modified based on investigator discretion. The duration of FST will be approximately 7 hours.

During the study, subjects will continue with their current diabetes regimen independent of the study devices. Subjects will be instructed by the investigational center that they are not to use the study devices (except for the CONTOUR™* study meter) for the management of their diabetes. The CONTOUR™* study meter may be used for treatment decisions and calibration of Guardian™ Sensor (3).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 14 - 75 years of age at time of screening
2. Subject has a clinical diagnosis of type 1 or 2 diabetes as determined via medical record or source documentation by an individual qualified to make a medical diagnosis
3. Subject has adequate venous access as assessed by investigator or appropriate staff
4. Subject is willing to follow the study procedures and willing to come to study visits

Exclusion Criteria:

1. Subject will not tolerate tape adhesive in the area of Guardian™ Sensor (3) placement as assessed by qualified individual.
2. Subject has any unresolved adverse skin condition in the area of study device or device placement (e.g., psoriasis, rash, Staphylococcus infection)
3. Subject is actively participating in an investigational study (drug or device) wherein they have received treatment from an investigational study (drug or device) in the last 2 weeks
4. Subject is female and has a positive pregnancy screening test
5. Females of child bearing age and who are sexually active should be excluded if they are not using a form of contraception deemed reliable by investigator
6. Subject is female and plans to become pregnant during the course of the study
7. Subject has a hematocrit (Hct) lower than the normal reference range
8. Subject may not be on the research staff of those performing this study

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, MD, Principal Investigator — Shanghai 6th People's Hospital; Xiaofeng Lv, MD, Principal Investigator — Seventh Medical Center of PLA Army General Hospital; Hong Li, MD, Principal Investigator — Sir Run Run Shaw Hospital
Locations (3):
- China (3):
  - The Seventh Medical Center of PLA General Hospital, Beijing
  - Sir Run Run Shaw Hospital, Hangzhou
  - Shanghai Sixth People's Hospital, Shanghai

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 72 subjects consented and enrolled in the overall study. Of the 72, 3 subjects failed screening, 3 subjects didn't utilize any Guardian™ Sensor (3) , 66 subjects utilized Guardian™ Sensor (3) and were considered to have started in the study.
Period: Overall Study
Arm/Group | Study Arm
Started | 66
Completed | 63
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Unsuccessful Procedure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Study Arm
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.67 (17.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han Chinese | 64
  Hui Chinese | 1
  Man Chinese | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.51 (3.61)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Guardian™ Sensor (3) Values That Are Within 20% Agreement of YSI
Description: Percentage of Guardian™ Sensor (3) Values that are within 20% agreement of Yellow Springs Instrument (YSI) plasma glucose values (±20 mg/dL (1.1 mmol/L) when reference blood glucose (YSI) less than or equal to (≤) 80 mg/dL (4.4 mmol/L) ) during YSI frequent sampling testing (FST) days.
Time Frame: 168 Hours
Population: A total of 63 subjects who had Guardian™ Sensor (3) inserted and had at least one paired Guardian™ Sensor (3) value and YSI measurement.
Measure: Mean (95% Confidence Interval); unit: percentage of paired readings
Arm/Group | Study Arm
Number analyzed (Participants) | 63
percentage of paired readings | 93.2 [92.1 to 94.4]

2. Primary Outcome: Consensus Error Grid Analysis of Mean Rate of Paired Sensor Values and YSI Values in Zone A+B
Description: A mean rate in Zone A+B of Consensus Error Grid between Guardian Sensor (3) values and YSI™* plasma glucose values during YSI™* FST days was evaluated. Consensus Error Grid (or Parkes error grid) compared the paired primary sensor and YSI reference glucose values. Zone A is defined in the Parkes error grid as the zone of "clinical accurate measurements with no effect on clinical action", Zone B as "altered clinical action with little or no effect on clinical outcome". Ideal situation is 100% in Zone A + B.
Time Frame: 168 Hours
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of paired readings
Arm/Group | Study Arm
Number analyzed (Participants) | 63
percentage of paired readings | 100 [100 to 100]

3. Primary Outcome: Clarke Error Grid Analysis of Mean Rate of Paired Sensor Values and YSI Values in Zone A+B
Description: A mean rate in Zone A+B of Clarke Error Grid between Guardian Sensor (3) values and YSI™* plasma glucose values during YSI™* FST days was evaluated. Clarke Error Grid compared the paired primary sensor and YSI reference glucose values. Zone A are "clinically accurate in that they would lead to clinically correct treatment decisions". Zone B "would lead to benign or no treatment". Ideal situation is 100% in Zone A + B.
Time Frame: 168 Hours
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of paired readings
Arm/Group | Study Arm
Number analyzed (Participants) | 63
percentage of paired readings | 99.8 [99.5 to 100]

4. Primary Outcome: Mean Absolute Relative Difference (MARD)
Description: Mean absolute relative difference (MARD) between Guardian Sensor (3) values and YSI™* plasma glucose values during YSI™* FST days was evaluated. MARD = Mean of ((Absolute difference of YSI reference and Sensor glucose values / YSI reference glucose values) * 100). Therefore, the unit of MARD is percentage (%). Note that results from multiple FST days were pooled together for reporting purpose.
Time Frame: 168 Hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of difference
Arm/Group | Study Arm
Number analyzed (Participants) | 63
percentage of difference | 8.11 (4.02)

ADVERSE EVENTS:
Time Frame: 7 days (from sensor insertion to end of study)
Arm/Group | Study Arm
All-Cause Mortality (participants affected / at risk) | 0/66
Serious Adverse Events (participants affected / at risk) | 0/66
Other Adverse Events (participants affected / at risk) | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/83/NCT03710083/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-14): https://cdn.clinicaltrials.gov/large-docs/83/NCT03710083/SAP_001.pdf